CLINICAL TRIAL: NCT03775200
Title: The Safety and Efficacy of Psilocybin in Participants With Treatment Resistant Depression
Acronym: P-TRD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: COMPASS Pathways (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COMP001
Record Dates: First submitted 2018-12-11; First posted 2018-12-13 (Actual); Results first posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Psilocybin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low dose (Experimental): Low dose Psilocybin
  Interventions: Drug: Psilocybin
- Medium dose (Experimental): Medium dose Psilocybin
  Interventions: Drug: Psilocybin
- High dose (Experimental): High dose Psilocybin
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — Dose-finding

SUMMARY:
The Safety and Efficacy of Psilocybin in Participants with Treatment Resistant Depression

DETAILED DESCRIPTION:
The Safety and Efficacy of Psilocybin in Participants with Treatment Resistant Depression - a dose-ranging study

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of TRD

Exclusion Criteria:

* Other comorbidities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-09-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (8):
  - Kadima Neuropsychiatry Institute, La Jolla, California
  - Altman Clinical and Translational Research Institute, University of California, San Diego, California
  - Stanford Department of Psychiatry, Stanford, California
  - Mood and Anxiety Disorders Program Emory University School of Medicine, Atlanta, Georgia
  - Ray Worthy Psychiatry LLC, New Orleans, Louisiana
  - Sheppard Pratt Health System, Baltimore, Maryland
  - New York State Psychiatric Institute, New York, New York
  - UT Center of Excellence on Mood Disorders, University of Texas Health Science Center, Houston, Texas
- Canada (2):
  - Canadian Rapid Treatment Centre of Excellence, Mississauga, Ontario
  - Centre for Addiction and Mental Health, Toronto, Ontario
- National Institute of Mental Health Czech Republic, Klecany, Czechia
- Enhed for Psykiatrisk Forskning, Psykiatrien i Aalborg, Aalborg, Denmark
- Charité - Universitätsmedizin Berlin, Department of Psychiatry and Psychotherapy, Campus Benjamin Franklin, Berlin, Germany
- Tallaght University Hospital, Dublin, Ireland
- Netherlands (3):
  - Groningen University Medical Centre, Groningen
  - Leiden University Medical Centre, Leiden
  - Utrecht University Medical Centre, Utrecht
- Unidade de Neuropsiquiatria, Centro Clinico Champalimaud, Lisbon, Portugal
- Spain (2):
  - Hospital de Dia Numancia, Barcelona
  - Institute Hospital del Mar of Medical Research (IMIM), Barcelona
- United Kingdom (5):
  - Clinical Research and Imaging Centre, Bristol, Avon
  - Wolfson Research Centre, Campus for Ageing and Vitality, Newcastle upon Tyne, Tyne and Wear
  - St. Pancras Clinical Research, London
  - Kings College London, Institute of Psychiatry, Psychology and Neurology, London
  - Greater Manchester Mental Health Foundation Trust, Manchester

REFERENCES:
- [Derived] Kirlic N, Atli M, Mistry S, Gold M, Goodwin GM. The Relationship Between Participant Pretreatment Clinical Presentation and the Quality of Psilocybin Experience: A Retrospective Analysis. J Clin Psychopharmacol. 2025 Dec 9. doi: 10.1097/JCP.0000000000002119. Online ahead of print. PMID 41362124
- [Derived] Goodwin GM, Aaronson ST, Alvarez O, Arden PC, Baker A, Bennett JC, Bird C, Blom RE, Brennan C, Brusch D, Burke L, Campbell-Coker K, Carhart-Harris R, Cattell J, Daniel A, DeBattista C, Dunlop BW, Eisen K, Feifel D, Forbes M, Haumann HM, Hellerstein DJ, Hoppe AI, Husain MI, Jelen LA, Kamphuis J, Kawasaki J, Kelly JR, Key RE, Kishon R, Knatz Peck S, Knight G, Koolen MHB, Lean M, Licht RW, Maples-Keller JL, Mars J, Marwood L, McElhiney MC, Miller TL, Mirow A, Mistry S, Mletzko-Crowe T, Modlin LN, Nielsen RE, Nielson EM, Offerhaus SR, O'Keane V, Palenicek T, Printz D, Rademaker MC, van Reemst A, Reinholdt F, Repantis D, Rucker J, Rudow S, Ruffell S, Rush AJ, Schoevers RA, Seynaeve M, Shao S, Soares JC, Somers M, Stansfield SC, Sterling D, Strockis A, Tsai J, Visser L, Wahba M, Williams S, Young AH, Ywema P, Zisook S, Malievskaia E. Single-Dose Psilocybin for a Treatment-Resistant Episode of Major Depression. N Engl J Med. 2022 Nov 3;387(18):1637-1648. doi: 10.1056/NEJMoa2206443. PMID 36322843
- [Derived] Kelly JR, Baker A, Babiker M, Burke L, Brennan C, O'Keane V. The psychedelic renaissance: the next trip for psychiatry? Ir J Psychol Med. 2022 Dec;39(4):335-339. doi: 10.1017/ipm.2019.39. Epub 2019 Sep 23. PMID 31543078

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient first visit: 1 March 2019 Last patients last visit: 27 September 2021
Groups:
- 25 mg COMP360 Psilocybin: 25 mg COMP360 Psilocybin
- 10 mg COMP360 Psilocybin: 10 mg COMP360 Psilocybin
- 1 mg COMP360 Psilocybin: 1 mg COMP360 Psilocybin
Period: Overall Study
Arm/Group | 25 mg COMP360 Psilocybin | 10 mg COMP360 Psilocybin | 1 mg COMP360 Psilocybin
Started | 79 | 75 | 79
Completed | 74 | 66 | 69
Not Completed | 5 | 9 | 10

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all randomised participants who received study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | 25 mg COMP360 Psilocybin | 10 mg COMP360 Psilocybin | 1 mg COMP360 Psilocybin | Total
Number analyzed (Participants) | 79 | 75 | 79 | 233
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 76 | 73 | 77 | 226
  >=65 years | 3 | 2 | 2 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at Screening
  years | 40.2 (12.19) | 40.6 (12.76) | 38.7 (11.71) | 39.8 (12.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 34 | 43 | 112
  Male | 44 | 41 | 36 | 121
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 4 | 3 | 5 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 0 | 1 | 5
  White | 70 | 72 | 73 | 215
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 2 | 2 | 2 | 6
  Netherlands | 17 | 16 | 17 | 50
  United States | 32 | 32 | 32 | 96
  Czechia | 3 | 2 | 2 | 7
  Ireland | 3 | 3 | 5 | 11
  Denmark | 3 | 2 | 3 | 8
  United Kingdom | 11 | 10 | 12 | 33
  Portugal | 1 | 0 | 1 | 2
  Germany | 2 | 2 | 0 | 4
  Spain | 5 | 6 | 5 | 16

OUTCOME MEASURES:

1. Primary Outcome: Montgomery Asberg Depression Rating Scale (MADRS) Change From Baseline to Week 3
Description: MADRS is a clinician-rated scale measuring depression symptom severity, consisting of 10 items, each scored from 0 (normal) to 6 (severe), for a total possible score of between 0 to 60; higher scores denote greater severity. Response >= 50% decrease and remission <= 10 total score.
Time Frame: Change from Baseline to Week 3
Population: The full analysis set includes all participants randomised who receive study drug and have at least 1 post-dose efficacy assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 25 mg COMP360 Psilocybin | 10 mg COMP360 Psilocybin | 1 mg COMP360 Psilocybin
Number analyzed (Participants) | 79 | 75 | 79
units on a scale | -12 (12.98) | -8.9 (10.94) | -6.8 (11.10)
Statistical Analysis 1: Comparison: 25 mg COMP360 Psilocybin vs 1 mg COMP360 Psilocybin; The primary analysis was the comparison between COMP360 (25 mg or 10 mg) versus COMP360 1 mg. The null hypothesis was that there was no difference in mean change from Baseline in MADRS total score at Week 3 for COMP360 25 mg or COMP360 10 mg versus COMP360 1 mg. The alternative hypothesis was that were was a difference in mean change from Baseline in MADRS total score at Week 3 for COMP360 25 mg or COMP360 10 mg versus COMP360 1 mg; Test type: Other — For this primary analysis, a sample size of 216 randomised participants (72:72:72) will provide 90% power at the alpha = 0.05 level to detect a 6-point difference in average MADRS total score between the optimal therapeutic dose of COMP360 and COMP360 1 mg, assuming the common standard deviation (SD) is 11.0; p < 0.05, Mixed Models Analysis; Hypothetical strategy estimand - missing not at random (MNAR) and missing at random (MAR) imputation for missing data; Least Mean Square Difference = -6.6, 95% CI 2-sided [-10.2 to -2.9], Standard Error of Mean 1.86 — LSM difference of COMP360 25 mg compared to COMP360 1 mg

2. Primary Outcome: MADRS Change From Baseline to Week 3, Sensitivity Analysis
Description: as for outcome 1
Time Frame: Change from Baseline to Week 3
Population: The per-protocol analysis set includes all participants in the Full Analysis Set who do not have a protocol deviation that is thought to significantly affect the integrity of the participant's efficacy data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 25 mg COMP360 Psilocybin | 10 mg COMP360 Psilocybin | 1 mg COMP360 Psilocybin
Number analyzed (Participants) | 77 | 65 | 68
units on a scale | -12 (12.98) | -8.9 (11.11) | -6.7 (11.18)
Statistical Analysis 1: Comparison: 25 mg COMP360 Psilocybin vs 1 mg COMP360 Psilocybin; Sensitivity analysis of the primary endpoint using the per-protocol analysis set; Test type: Other; p < 0.05, Mixed Models Analysis; Hypothetical strategy estimand - MNAR and MAR imputation for missing data; Least Mean Square Difference = -5.6, 95% CI 2-sided [-9.4 to -1.8], Standard Error of Mean 1.93

ADVERSE EVENTS:
Time Frame: Up to 12 Weeks
Description: The Safety Analysis Set included all randomised participants who received study drug.
Arm/Group | 25 mg COMP360 Psilocybin | 10 mg COMP360 Psilocybin | 1 mg COMP360 Psilocybin
All-Cause Mortality (participants affected / at risk) | 0/79 | 0/75 | 0/79
Serious Adverse Events (participants affected / at risk) | 5/79 | 6/75 | 1/79
Other Adverse Events (participants affected / at risk) | 60/79 | 51/75 | 50/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 25 mg COMP360 Psilocybin (N=79) | 10 mg COMP360 Psilocybin (N=75) | 1 mg COMP360 Psilocybin (N=79)
Drug withdrawal syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0)
Suicidal behaviour (Psychiatric disorders) | 3 (3) | 0 (0) | 0 (0)
Intentional self-injury (Psychiatric disorders) | 2 (2) | 2 (2) | 1 (2)
Adjustment disorder with anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Adjustment disorder with mixed anxiety and depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 2 (2) | 2 (3) | 0 (0)
Hospitalisation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 25 mg COMP360 Psilocybin (N=79) | 10 mg COMP360 Psilocybin (N=75) | 1 mg COMP360 Psilocybin (N=79)
Nausea (Gastrointestinal disorders) | 18 (19) | 7 (7) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 4 (4) | 2 (2) | 1 (1)
Fatigue (General disorders) | 12 (12) | 5 (5) | 7 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 0 (0) | 3 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 27 (34) | 16 (22) | 20 (30)
Dizziness (Nervous system disorders) | 6 (6) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 3 (3) | 4 (4) | 1 (1)
Insomnia (Psychiatric disorders) | 8 (8) | 11 (11) | 14 (16)
Anxiety (Psychiatric disorders) | 7 (7) | 13 (16) | 3 (3)
Depression (Psychiatric disorders) | 4 (4) | 5 (5) | 5 (5)
Euphoric mood (Psychiatric disorders) | 4 (4) | 5 (5) | 4 (5)
Depressed mood (Psychiatric disorders) | 3 (3) | 5 (5) | 4 (5)
Suicidal ideation (Psychiatric disorders) | 5 (5) | 3 (3) | 4 (5)
Mood altered (Psychiatric disorders) | 7 (8) | 3 (3) | 1 (1)
Irritability (Psychiatric disorders) | 4 (4) | 2 (2) | 1 (1)
Panic reaction (Psychiatric disorders) | 4 (4) | 1 (1) | 1 (1)
Thinking abnormal (Psychiatric disorders) | 0 (0) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-07-22): https://cdn.clinicaltrials.gov/large-docs/00/NCT03775200/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-26): https://cdn.clinicaltrials.gov/large-docs/00/NCT03775200/SAP_001.pdf